CLINICAL TRIAL: NCT06865599
Title: Evaluation of the Effectiveness of a Program on Breastfeeding for Medical Interns Assiut University
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Albatoul Nageh Fouly, demonstrator at public health department ,Assiut university, Assiut University
Other Study IDs: Breastfeeding medical interns
Record Dates: First submitted 2025-03-06; First posted 2025-03-10 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: Intern doctors integrated system (5+2) Intern doctors graduated from Assiut University September 2024.

SUMMARY:
The WHO and UNICEF advocate for infants to start nursing within the first hour post-birth and to be exclusively breastfed for the first six months of life. Commencing at six months of age, children should start the consumption of safe and sufficient supplemental meals while maintaining breastfeeding for up to two years or longer (WHO), 2025) . Abd El Khalek et al. assessed the impact of instructional guidelines on 100 pregnant women at South Valley University Hospital. Initially, most had poor knowledge, negative attitudes, and inadequate practices. After one month of guidelines implementation, significant improvements in women awareness regrading breastfeeding were observed . Bahaa et al. reported that breastfeeding is a critical concern for the entire community. Their study assessed the knowledge and practices of 261 lactating mothers at Awlad Saqr Center Al Sharkia governate.

Findings showed that 73.2% practiced EBF, while only 45.2% had sufficient knowledge. Intentions for EBF for six months were high (86.2%). The study concluded that despite acceptable EBF rates, knowledge gaps remain, highlighting the need to enhance counseling services during antenatal and postnatal care .

One of the best ways to improve the survival and condition of newborns is breastfeeding . Ensuring ideal breastfeeding habits depends significantly on the encouragement and assistance of healthcare workers, especially physicians. A program on breastfeeding for medical interns is crucial to find gaps and helping to enhance medical support and education within the healthcare system. The overall aim is to evaluate the effectiveness of an educational program on breastfeeding for the medical intern at Assiut University.

Specific objectives:

1. Evaluation of the knowledge regarding breastfeeding for medical interns.
2. Implementing an educational program based on the UNICEF Baby-Friendly Initiative for the medical intern.
3. Measuring the effectiveness of the educational program on breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

Unmarried intern doctors Both male and female intern doctors Intern doctors integrated system (5+2) Intern doctors graduated from Assiut University September 2024

Exclusion Criteria:

* Intern doctors who have previous health education sessions about breastfeeding. Intern doctors

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Intern doctors integrated system (5+2) graduated from Assiut University September 2024
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of the program | baseline
  Success rate of the program by calculating mean and standard deviation of total knowledge scores pre and post the educational program